CLINICAL TRIAL: NCT05625191
Title: Defining Clinically Important Differences in Cepstral and Spectral Measures in Individuals With and Without Phonotrauma
Brief Title: Patients With and Without Phonotrauma
Status: Recruiting | Type: Observational
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Laura Toles, PhD, Assistant Professor, University of Texas Southwestern Medical Center
Other Study IDs: STU-2022-0655
Record Dates: First submitted 2022-11-02; First posted 2022-11-22 (Actual); Last update posted 2025-07-30 (Actual); Status verified 2025-07

CONDITIONS: Phonotrauma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Control Group- Without Phonotrauma: Videoendoscopy and acoustic recordings using a head-mounted microphone with a voice-specialized SLP for participants without voice disorders, acoustic recordings will involve the five repetitions of three vowels (/ɑ, i, u/) and a standard reading passage (Rainbow Passage) in three voice conditions (breathy, typical, and pressed). For all participants, high-speed videoendoscopy and simultaneous acoustic recording will occur on one repetition of a sustained /i/ in each requested condition.
  Interventions: Diagnostic Test: Acoustic voice analysis
- Patients Diagnosed with Phonotrauma: Videoendoscopy and acoustic recordings using a head-mounted microphone with a voice-specialized SLP for Participants who have a diagnosis of phonotrauma will be instructed to produce five repetitions of the same three vowels but in only two conditions: typical voice and "resonant" voice following stimulability assessment and with cues. They will be instructed to maintain relatively consistent volume and pitch across conditions. For all participants, high-speed videoendoscopy and simultaneous acoustic recording will occur on one repetition of a sustained /i/ in each requested condition.
  Interventions: Diagnostic Test: High-speed videoendoscopy

INTERVENTIONS:
Diagnostic Test: Acoustic voice analysis — Acoustic recordings will involve the five repetitions of three vowels (/ɑ, i, u/) and a standard reading passage (Rainbow Passage) in different voice conditions. Control participants will produce voice in breathy, typical, and pressed conditions. Patient participants will produce voice in typical production and in a resonant voice production. High-speed videoendoscopy and simultaneous acoustic recording will occur on one repetition of a sustained /i/ in each requested condition. Data will be collected using a head-mounted microphone.
  Groups: Control Group- Without Phonotrauma
Diagnostic Test: High-speed videoendoscopy — High-speed videoendoscopy will occur on one repetition of a sustained /i/ in each requested condition. Exams will be recorded using the Phantom V311 high-speed camera (Vision Research, Wayne, NJ) connected to a Storz 70° rigid laryngoscope using a 400 Watt Xenon light source (Titan 400E).
  Groups: Patients Diagnosed with Phonotrauma

SUMMARY:
There is a substantial need to identify objective measures associated with hyperadduction of the vocal folds to recognize those at higher risk of developing phonotrauma so that risk mitigation strategies can be implemented before phonotrauma develops. The overall objective of this proposed project is to investigate the sensitivity and direction of change in cepstral peak prominence (CPP) and the magnitude difference between the first two harmonics of the voice spectrum (H1-H2) in response to varied phonation patterns, which will be addressed using the following two aims:

Aim 1: Determine how CPP and H1-H2 change as a function of using pressed voice production in individuals without laryngeal pathology.

Aim 2: Examine the sensitivity (minimally detectable change) and responsiveness (minimal clinically important difference) of CPP and H1-H2 to detect changes in different voice production conditions.

ELIGIBILITY:
Control Group:

Inclusion Criteria:

1. 18-65 years of age (to avoid confounding physiological factors related to puberty or presbyphonia)
2. No history of or current voice disorder
3. Auditory perceptual presentation globally within functional limits (as determined by a voice specialized SLP).

Exclusion Criteria:

1. Atypical auditory-perceptual voice presentation
2. History of voice disorder or laryngeal surgery.

Patient Group:

Inclusion Criteria:

1. Diagnosed with phonotrauma (i.e., vocal fold nodules, vocal fold polyp, vocal fold pseudocyst, mid-fold edema) by a laryngologist.
2. 18-65 years of age

Exclusion Criteria:

1. Diagnosis of voice disorder not related to phonotrauma (e.g., vocal fold immobility, laryngeal dystonia, primary muscle tension dysphonia, etc.)
2. Previous history of laryngeal surgery or voice therapy (to avoid confounding effects of previous treatment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients (18-65 years of age) with a diagnosis of phonotrauma will be recruited from the laryngology clinics at UTSW Voice Center. All patients who are diagnosed with phonotraumatic vocal fold lesions (including vocal fold nodules, phonotraumatic polyps, mid-fold edema, and pseudocysts) will be referred for enrollment. Individuals without phonotrauma (18-65 years of age) will be recruited for the control group.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Cepstral Peak Prominence | 1 year
  Cepstral peak prominence is a measure of the periodic energy of the acoustic voice signal.
The difference between the first and second harmonic (H1-H2) | 1 year
  H1-H2 is a spectral measure derived from the acoustic voice signal that correlates with glottal configuration.
Average closing velocity | 1 year
  Vocal fold closing phase velocity averaged across 100 vibratory cycles

CONTACTS AND LOCATIONS:
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

REFERENCES:
- [Background] Hillman RE, Stepp CE, Van Stan JH, Zanartu M, Mehta DD. An Updated Theoretical Framework for Vocal Hyperfunction. Am J Speech Lang Pathol. 2020 Nov 12;29(4):2254-2260. doi: 10.1044/2020_AJSLP-20-00104. Epub 2020 Oct 2. PMID 33007164
- [Background] Verdolini K, Hess MM, Titze IR, Bierhals W, Gross M. Investigation of vocal fold impact stress in human subjects. J Voice. 1999 Jun;13(2):184-202. doi: 10.1016/s0892-1997(99)80022-8. PMID 10442749
- [Background] Klatt DH, Klatt LC. Analysis, synthesis, and perception of voice quality variations among female and male talkers. J Acoust Soc Am. 1990 Feb;87(2):820-57. doi: 10.1121/1.398894. PMID 2137837
- [Background] Awan SN, Roy N, Jette ME, Meltzner GS, Hillman RE. Quantifying dysphonia severity using a spectral/cepstral-based acoustic index: Comparisons with auditory-perceptual judgements from the CAPE-V. Clin Linguist Phon. 2010 Sep;24(9):742-58. doi: 10.3109/02699206.2010.492446. PMID 20687828
- [Background] Murton O, Hillman R, Mehta D. Cepstral Peak Prominence Values for Clinical Voice Evaluation. Am J Speech Lang Pathol. 2020 Aug 4;29(3):1596-1607. doi: 10.1044/2020_AJSLP-20-00001. Epub 2020 Jul 13. PMID 32658592
- [Background] Toles LE, Ortiz AJ, Marks KL, Burns JA, Hron T, Van Stan JH, Mehta DD, Hillman RE. Differences Between Female Singers With Phonotrauma and Vocally Healthy Matched Controls in Singing and Speaking Voice Use During 1 Week of Ambulatory Monitoring. Am J Speech Lang Pathol. 2021 Jan 27;30(1):199-209. doi: 10.1044/2020_AJSLP-20-00227. Epub 2021 Jan 20. PMID 33472007